CLINICAL TRIAL: NCT06639386
Title: Examining Underlying Factors and Root Cause of Successful Evidence Based Interventions (EBIs) Among Historically Marginalized Racial and Ethnic Groups Using the Consolidated Framework for Implementation Research (CFIR)
Brief Title: Vaccine Confidence Study Among Historically Marginalized Racial and Ethnic Groups
Status: Recruiting | Type: Observational
Sponsor: Boston Medical Center (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: H-44825
Record Dates: First submitted 2024-10-10; First posted 2024-10-15 (Actual); Last update posted 2025-07-17 (Actual); Status verified 2025-07

CONDITIONS: Vaccine Hesitancy; Vaccine Refusal
Keywords: Vaccine confidence; Marginalized populations; MMR vaccine; RSV vaccine
MeSH Terms: conditions — Vaccination Hesitancy; Vaccination Refusal

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Parents of children 12-24 months: 30 birthing parents and their 12-24 month old infants will be enrolled into the study. Study activities (enrollment and interviews) can be conducted with participants in English, Haitian Creole, or Spanish.
- Clinicians: 35 clinicians at BMC will be recruited to participate in anonymous, one-time interviews. The sample will include 20 Community Health Workers, 10 pediatric/family Medicine clinicians, and 5 Obstetricians. Recruitment will focus on clinicians who have a history of successful vaccine-specific Evidence-Based Interventions (EBIs) beyond BMC and its affiliated CHCs.
- Evidence Based Intervention (EBI) Experts: 15 EBI Experts will be identified from a literature review of published peer-review articles in the fields of vaccine EBIs, implementation science, and prenatal genetic counseling.

SUMMARY:
Achieving optimal vaccination rates is vital for protecting the health and well-being of all individuals. This specific study focuses on the MMR and RSV vaccines in pregnancy and early childhood, which have been shown to reduce RSV and MMR-related illnesses, hospitalizations, and deaths. Efforts to improve vaccination rates have not been equally effective across the entire population; this has resulted in poorer outcomes from interventions for certain populations who are vaccine-hesitant.

This study seeks to understand how to best increase vaccine confidence in marginalized populations. To do this, the investigators will interview parents of children who receive care at Boston Medical Center (BMC), Community Health Workers and other Clinical providers at BMC, leading experts in the fields of vaccine confidence and implementation science, and key public health stakeholders/officials.

ELIGIBILITY:
Inclusion Criteria:

Parent and child-

* The birthing parent of any age of a child (aged 12-24 months) who receives primary care at Boston Medical Center
* A birthing parent who is registered as a patient at Boston Medical Center
* The birthing parent must have been pregnant between the months of October and February (RSV season)
* The birthing parent must be comfortable completing an interview in English, Spanish, or Haitian Creole.

Clinician

* Clinical provider (including Community Health Workers, Physicians, Physician Assistants and Nurse Practitioners) aged 18+ years at Boston Medical Center within Pediatrics, Family Medicine, or OB/GYN. These clinicians will have been involved in past or current successful vaccine-specific Evidence Based Interventions (EBI) beyond BMC and its affiliated Community Health Center (CHC).

EBI Expert

* Content experts (aged 18+ years) in the areas of Implementation Science, Vaccine-specific EBIs, and Prenatal genetic counseling

Exclusion Criteria:

* Clinical provider (including Community Health Workers, Physicians, Physician Assistants and Nurse Practitioners) at NON-BMC clinic/Community Health Center
* Content experts - NON-Vaccine evidence based interventions (EBIs)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The population of 30 adult parents of children 12-24 months will be identified from a clinical database of patients registered at Boston Medical Center (BMC).
  The 35 clinicians will be identified from from Pediatrics, Family Medicine, or obstetrics and gynecology (OB/GYN) at BMC. The sample will include 20 Community Health Workers, 10 pediatric/family Medicine clinicians, and 5 Obstetricians. Recruitment will focus on clinicians who have a history of successful vaccine-specific Evidence-Based Interventions (EBIs) beyond BMC and its affiliated CHCs.
  The 15 evidence based interventions (EBI) experts will be identified from a review of published peer-review articles in the fields of vaccine EBIs, implementation science, and prenatal genetic counseling.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2025-01-31 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Vaccine confidence from the parents' perspective | 12 months
  Interviews will be conducted with parents and themes will be abstracted that relate to vaccine confidence. Counts of participants for each theme will be reported.
Vaccine confidence from the clinicians' perspective | 12 months
  Interviews will be conducted with clinicians and themes will be abstracted that relate to vaccine confidence. Counts of participants for each theme will be reported.
Vaccine confidence from the EBI Experts' perspective | 12 months
  Interviews will be conducted with EBI experts and themes will be abstracted that relate to vaccine confidence. Counts of participants for each theme will be reported.

CONTACTS AND LOCATIONS:
Overall Officials: Michelle Stransky, PhD, Principal Investigator — Boston Medical Center, Pediatrics
Locations (1):
- Boston Medical Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Undecided